CLINICAL TRIAL: NCT07395713
Title: The Effectiveness of Using Artificial Intelligence (Chat GPT) in Cardiac Assessment During Anesthesia Examination of Preoperative Cases
Brief Title: The Predictability of the Necessity for Cardiology Consultation in Patients Scheduled for Non-Cardiac Surgery Using Artificial Intelligence Models in Preoperative Anesthesia Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, eralp çevikkalp, associate professor, Bursa City Hospital
Other Study IDs: Bursa Şehir Hastanesi
Record Dates: First submitted 2025-12-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: USE OF ARTIFICIAL INTELLIGENCE IN ANESTHESIA; PREOPERATIVE CARDIOLOGY CONSULTATION REQUIREMENT
Keywords: THE ROLE OF ARTIFICIAL INTELLIGENCE IN ANESTHESIA; ARTIFICIAL INTELLIGENCE IN CONSULTATION NEEDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient scenarios were presented to different AI models (ChatGPT 4.5, ChatGPT 5, Copilot, Deepseek, Grok, Claude, Gemini Flash, Gemini Pro) with and without prompts. — Responses:
  Compared with expert opinion according to the ESC 2024 guidelines
  Evaluated using the Ateşman readability score and the Global Quality Scale (GQS)

SUMMARY:
Structured Summary Title

Predictability of Cardiology Consultation Requirement in Patients Undergoing Non-Cardiac Surgery Using Artificial Intelligence Models

Background

Preoperative cardiac risk assessment is essential for minimizing perioperative morbidity and mortality in patients undergoing non-cardiac surgery. Cardiology consultations are often requested to assess surgical eligibility and reduce complication risks. However, unnecessary consultations may contribute to inefficient healthcare resource utilization and procedural delays.

Recent advances in artificial intelligence, particularly large language models, have demonstrated potential in clinical decision support systems. The European Society of Cardiology (ESC) 2024 guidelines provide a structured framework for evaluating perioperative cardiac risk. This study aims to investigate whether AI-based models can assist in predicting the need for cardiology consultation and to examine the effect of prompted versus non-prompted input formats on AI recommendations.

Study Design

Prospective, observational, comparative study.

Ethical Approval

The study has been approved by the Bursa City Hospital Ethics Committee and will be conducted in accordance with the Declaration of Helsinki.

Sample Size

Sample size was calculated using G*Power software based on anticipated effect size and statistical power requirements.

Participants

Inclusion Criteria:

Adults aged 18 years or older

ASA physical status I-IV

Scheduled for non-cardiac surgery

Evaluated by anesthesia residents with less than two years of clinical experience

Exclusion Criteria:

Pediatric patients

Patients declining participation

Incomplete clinical data

Data Collection

The following patient data will be recorded:

Demographics (age, sex, BMI)

Medical history (comorbidities, medication use, allergies, substance use)

Functional capacity (METs score)

ECG findings

Chest radiography findings

Planned surgical procedure characteristics

AI Model Evaluation

Multiple AI language models will be tested using standardized patient scenarios. Each scenario will be presented in two formats:

Prompted format:

"You are a 10-year experienced anesthesiologist. According to ESC 2024 guidelines, evaluate whether this patient requires cardiology consultation."

Non-prompted format:

"Evaluate whether this patient requires cardiology consultation."

AI recommendations will not influence clinical decision-making.

Outcome Measures

Primary and secondary analyses will include:

Agreement between AI recommendations and expert anesthesiologist evaluations

Readability of AI-generated responses

Quality assessment of responses

Classification performance comparisons across models

Statistical Analysis

Statistical analyses will be performed using appropriate comparative and agreement tests. Readability and quality scores will be analyzed using non-parametric methods where applicable. ROC analysis will be used to assess classification ability. A significance level of p < 0.05 will be applied.

Study Objective

The objective of this study is to explore the feasibility of AI-assisted decision support systems in predicting cardiology consultation requirements and to evaluate whether prompt engineering influences AI performance.

DETAILED DESCRIPTION:
Structured Summary Title

Predictability of Cardiology Consultation Requirement in Patients Undergoing Non-Cardiac Surgery Using Artificial Intelligence Models

Background

Preoperative cardiac risk assessment is essential for minimizing perioperative morbidity and mortality in patients undergoing non-cardiac surgery. Cardiology consultations are often requested to assess surgical eligibility and reduce complication risks. However, unnecessary consultations may contribute to inefficient healthcare resource utilization and procedural delays.

Recent advances in artificial intelligence, particularly large language models, have demonstrated potential in clinical decision support systems. The European Society of Cardiology (ESC) 2024 guidelines provide a structured framework for evaluating perioperative cardiac risk. This study aims to investigate whether AI-based models can assist in predicting the need for cardiology consultation and to examine the effect of prompted versus non-prompted input formats on AI recommendations.

Study Design

Prospective, observational, comparative study.

Ethical Approval

The study has been approved by the Bursa City Hospital Ethics Committee and will be conducted in accordance with the Declaration of Helsinki.

Sample Size

Sample size was calculated using G*Power software based on anticipated effect size and statistical power requirements.

Participants

Inclusion Criteria:

Adults aged 18 years or older

ASA physical status I-IV

Scheduled for non-cardiac surgery

Evaluated by anesthesia residents with less than two years of clinical experience

Exclusion Criteria:

Pediatric patients

Patients declining participation

Incomplete clinical data

Data Collection

The following patient data will be recorded:

Demographics (age, sex, BMI)

Medical history (comorbidities, medication use, allergies, substance use)

Functional capacity (METs score)

ECG findings

Chest radiography findings

Planned surgical procedure characteristics

AI Model Evaluation

Multiple AI language models will be tested using standardized patient scenarios. Each scenario will be presented in two formats:

Prompted format:

"You are a 10-year experienced anesthesiologist. According to ESC 2024 guidelines, evaluate whether this patient requires cardiology consultation."

Non-prompted format:

"Evaluate whether this patient requires cardiology consultation."

AI recommendations will not influence clinical decision-making.

Outcome Measures

Primary and secondary analyses will include:

Agreement between AI recommendations and expert anesthesiologist evaluations

Readability of AI-generated responses

Quality assessment of responses

Classification performance comparisons across models

Statistical Analysis

Statistical analyses will be performed using appropriate comparative and agreement tests. Readability and quality scores will be analyzed using non-parametric methods where applicable. ROC analysis will be used to assess classification ability. A significance level of p < 0.05 will be applied.

Study Objective

The objective of this study is to explore the feasibility of AI-assisted decision support systems in predicting cardiology consultation requirements and to evaluate whether prompt engineering influences AI performance.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older

ASA physical status classification I-IV

Scheduled for non-cardiac surgery

Patients evaluated preoperatively by anesthesia residents with less than two years of clinical experience

Availability of complete clinical data including medical history, ECG findings, and chest radiography

Ability to provide informed consent

Exclusion Criteria:

Patients younger than 18 years of age

Patients undergoing cardiac surgery

Patients with incomplete clinical data

Patients who declined participation

Emergency surgery cases

Patients unable to undergo standard preoperative evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted with the participation of patients who will be referred to cardiology following an examination at the anesthesia clinic prior to undergoing non-cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Agreement Between AI Model Recommendations and Expert Anesthesiologist Decision Regarding Cardiology Consultation Requirement | At baseline preoperative evaluation (Day 1)
  The level of agreement between artificial intelligence model recommendations and expert anesthesiologist evaluations for cardiology consultation necessity will be assessed using Cohen's Kappa coefficient based on ESC 2024 guidelines.

OTHER OUTCOMES:
Readability of AI-Generated Responses | Immediately after AI-generated response evaluation (Day 1)
  The readability of AI-generated responses will be assessed using the Ateşman Readability Index to determine clarity and comprehensibility of consultation recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: eralp çevikkalp, Principal Investigator — bursa şehir hastanesi
Locations (1):
- Bursa Şehir Hastanesi, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to our commitment to patient rights, data privacy, and the consent form

REFERENCES:
- [Background] 1.M. Graeßner et al., "Enabling personalized perioperative risk prediction by using a machinelearning model based on preoperative data," Scientific Reports, vol. 13, no. 1, May 2023, doi: 10.1038/s41598-023-33981-8. 2.B. Choi et al., "Prediction Model for 30-Day Mortality after Non-Cardiac Surgery Using MachineLearning Techniques Based on Preoperative Evaluation of Electronic Medical Records," Journal of Clinical Medicine, vol. 11, no. 21, p. 6487, Nov. 2022, doi: 10.3390/jcm11216487. 3.M. Vine et al., "Innovative approaches to preoperative care including feasibility, efficacy, and ethical implications: a narrative review," AME Surgical Journal, vol. 4. AME Publishing Company, p. 1, Feb. 01, 2024. doi: 10.21037/asj-23-41. 4.P. Chung, C. T. Fong, A. M. Walters, N. Aghaeepour, M. Yetişgen, and V. N. O'Reilly-Shah, "Large Language Model Capabilities in Perioperative Risk Prediction and Prognostication," JAMA Surgery, vol. 159, no. 8, American Medical Association, p. 928, Jun. 05, 2024. doi: 10.1001/jamasurg.2024.1621 5.T. Yurttas, R. Hidvegi, and M. Filipovic, "Biomarker-Based Preoperative Risk Stratification for Patients Undergoing Non-Cardiac Surgery," Journal of Clinical Medicine, vol. 9, no. 2, p. 351, Jan. 2020, doi: 10.3390/jcm9020351 6.J. Stones and D. Yates, "Clinical risk assessment tools in anaesthesia," BJA Education, vol. 19, no. 2. Elsevier BV, p. 47, Dec. 15, 2018. doi: 10.1016/j.bjae.2018.09.009. 7. Engineering as an Important Emerging Skill for Medical Professionals: Tutorial. J Med Internet Res. 2023 Oct 4;25:e50638. doi: 10.2196/50638. PMID: 37792434; PMCID: PMC10585440. 8. ATEŞMAN, Ender. (1997). Türkçe'de okunabilirliğin Ölçülmesi. A.Ü. Tömer Dil Dergisi, sayı:58,s.171174. 9. Coskun B, Ocakoglu G, Yetemen M, Kaygisiz O. Can ChatGPT, an Artificial Intelligence Language Model, Provide Accurate and High-quality Patient Information on Prostate Cancer? Urology. 2023 Oct;180:35-58. doi: 10.1016/j.urology.2023.05.040. Epub 2023 Jul 4. PMID: 37406

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-12-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT07395713/SAP_000.pdf